CLINICAL TRIAL: NCT03526666
Title: Collection of Peripheral Blood From Patients With Myelodysplastic Syndrome, Acute Myeloid Leukemia, or Chronic Myelomonocytic Leukemia for Measuring Baseline Ascorbic Acid Levels and Future Epigenetic Cancer Research
Brief Title: Ascorbic Acid Levels in MDS, AML, and CMML Patients
Status: Completed | Type: Observational
Sponsor: Van Andel Research Institute (Other)
Responsible Party: Principal Investigator, Peter Jones, Cheif Scientific Officer, Van Andel Research Institute
Other Study IDs: 17022
Record Dates: First submitted 2018-05-03; First posted 2018-05-16 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-09

CONDITIONS: Myelodysplastic Syndromes; Acute Myeloid Leukemia; Chronic Myelomonocytic Leukemia; MDS; AML; CMML
Keywords: Vitamin C; Ascorbic Acid; Epigenetics; 5-hydroxymethylcytosine; 5-methylcytosine
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Plasma with ascorbic acid redox analysis prep (additive: MPA solution, 10 % meta-phosphoric acid w/v containing 2 mM Na2EDTA)
  2. Plasma
  3. Buffy coat pellet
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AML, MDS, and CMML patients: Patients with a diagnosis of acute myeloid leukemia (AML), myelodysplastic syndrome (MDS), or chronic myelomonocytic leukemia (CMML).
  Interventions: Other: Peripheral blood collection

INTERVENTIONS:
Other: Peripheral blood collection — Peripheral blood collection for the measurement of ascorbic acid levels and banking of plasma and buffy coat for future resrearch.

SUMMARY:
This study is a non-interventional, specimen collection translational study to evaluate vitamin C levels in the peripheral blood of Acute Myeloid Leukemia (AML), Myelodysplastic Syndrome (MDS), or Chronic Myelomonocytic Leukemia (CMML) patients.

DETAILED DESCRIPTION:
It has previously been established that hematological cancer patients with myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML) often exhibit severe vitamin C deficiency from a cohort of patients in Copenhagen. In this study, the investigators aim to determine if those results are conserved in another population/geographical location.

ELIGIBILITY:
Inclusion Criteria:

* Patients actively receiving treatment for acute myeloid leukemia (AML), myelodysplastic syndrome (MDS), or chronic myelomonocytic leukemia (CMML).
* Patients diagnosed with AML, MDS, or CMML and are treatment naïve.
* Patients who are 18 years old or older.

Exclusion Criteria:

* Patients deemed as too ill to participate as determined by the clinical investigator.
* Non-English speaking patients
* Patients unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen in hematology/oncology clinics in Grand Rapids, MI
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Peripheral blood ascorbic acid levels | 1 year
  The level of ascorbic acid

SECONDARY OUTCOMES:
Evaluation of human endogenous retroviral sequences (HERVs) expression | 1 year
Evaluation of 5-methylcitosine (5-mC) and 5-hydroxymethylcytosine (5-hmC) levels | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Peter Jones, Ph.D., D.Sc., Principal Investigator — Van Andel Research Institute
Locations (2):
- United States (2):
  - Cancer and Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - Metro Health - University of Michigan Health, Wyoming, Michigan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gillberg L, Orskov AD, Liu M, Harslof LBS, Jones PA, Gronbaek K. Vitamin C - A new player in regulation of the cancer epigenome. Semin Cancer Biol. 2018 Aug;51:59-67. doi: 10.1016/j.semcancer.2017.11.001. Epub 2017 Nov 2. PMID 29102482
- [Background] Liu M, Ohtani H, Zhou W, Orskov AD, Charlet J, Zhang YW, Shen H, Baylin SB, Liang G, Gronbaek K, Jones PA. Vitamin C increases viral mimicry induced by 5-aza-2'-deoxycytidine. Proc Natl Acad Sci U S A. 2016 Sep 13;113(37):10238-44. doi: 10.1073/pnas.1612262113. Epub 2016 Aug 29. PMID 27573823

DOCUMENTS (1):
  • Study Protocol (2018-02-09): https://cdn.clinicaltrials.gov/large-docs/66/NCT03526666/Prot_000.pdf